CLINICAL TRIAL: NCT01490424
Title: Association Between TREM-1 Gene Polymorphisms and Prognosis in Sepsis Patient
Brief Title: TREM-1 Gene Polymorphisms
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Other Study IDs: 20111013-009（2）; 2009BAI86B03 (Other Grant/Funding Number: Chinese National Science & Technology Pillar Program)
Record Dates: First submitted 2011-12-12; First posted 2011-12-13 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Sepsis
Keywords: TREM-1;; SNPs;; prognosis; control（normal person）
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- sepsis: SIRS plus inflammation
- Control: normal person under medical examination

SUMMARY:
Triggering receptor expressed on myeloid cells-1 (TREM-1) is a cell surface receptor expressed on neutrophils and monocytes. TREM-1 acts to amplify inflammation and serves as a critical mediator of inflammatory response in the context of sepsis. Blocking of TREM-1 can protect against sepsis in mice. This study was designed to investigate whether TREM-1 genomic variations were associated with the prognosis of sepsis. We sequenced 30 sepsis patients with TREM-1 gene of four exons by PCR sequencing. When analyzing the results of sequencing, we found two gene polymorphisms located in exon-2 and exon-4, respectively. Compare with the NCBI dbSNP and Hapmap database, one polymorphisms located in exon-2 is non-synonymous variation rs2234237（Ser25Thr）, the other one located in exon-4 is synonymous variation rs2234246. Two common polymorphisms (rs2234237,rs2234246) within the TREM-1 gene were detected in 80 patients with severe sepsis and in 80 healthy control subjects. This study was explored that whether or not polymorphisms detected within the TREM-1 gene may play a major role in the predisposition to prognosis of sepsis in a Chinese Han cohort.

ELIGIBILITY:
Inclusion Criteria:

* Sepsis met the criteria recommended by 1991 ACCP/SCCM Joint Meeting and by the diagnostic criteria developed at the 2001 International Sepsis Definition Conference.

Exclusion Criteria:

* (1) younger than 18 years of age; (2) acquired immunodeficiency syndrome; (3) reduced polymorphonuclear granulocyte counts (< 500 μL-1); (4) died within 24h after admission into the ICU, or refused to participate in the study, or declined treatment during the period of observation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All subjects were selected from among inpatients who were hospitalized between September 2009 and October 2011 in the Respiratory ICU, Surgical ICU, and Emergency ICU, Chinese People's Liberation Army (CPLA) General Hospital.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2010-05; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Patients Outcome | 28 days
  The survival time of patients more than 28days is defined as survival. The survival time of patients less than 28days is defined as death

CONTACTS AND LOCATIONS:
Overall Officials: Lixin Xie, MD, Study Director — Respiratory Disease Department of chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Su L, Liu C, Li C, Jiang Z, Xiao K, Zhang X, Li M, Yan P, Feng D, Xie L. Dynamic changes in serum soluble triggering receptor expressed on myeloid cells-1 (sTREM-1) and its gene polymorphisms are associated with sepsis prognosis. Inflammation. 2012 Dec;35(6):1833-43. doi: 10.1007/s10753-012-9504-z. PMID 22798017